CLINICAL TRIAL: NCT05284110
Title: Breaking up Sedentary Time in Rheumatoid Arthritis: Effects on Vascular Function
Brief Title: Breaking up Sedentary Time in Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BRAKETIME
Record Dates: First submitted 2022-02-24; First posted 2022-03-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis; Sedentary Behavior; Endothelial Dysfunction
Keywords: physical activity; rheumatic diseases; vascular function
MeSH Terms: conditions — Arthritis, Rheumatoid; Sedentary Behavior; Motor Activity; Rheumatic Diseases | interventions — Exercise; Walking

STUDY DESIGN:
Intervention Model Description: Participants with rheumatoid arthritis will attend the laboratory at Liverpool John Moores University on 2 occasions. During these visits, they will be submitted to the intervention or the control and will also undertake a series vascular tests prior- and post-intervention/control.
Who Masked: Outcomes Assessor
Masking Description: The researcher who will perform the vascular analysis will be blinded to the allocation order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking breaks (WALK) (Experimental): During this session, participants will be requested to remain seated during 4 hours, but the sitting will be interrupted every 30 min with a 3-min light-intensity walking.
  Interventions: Behavioral: Physical activity
- Prolonged sitting (SIT) (No Intervention): During this session, participants be requested to remain seated during 4 uninterrupted hours (excepted for visiting the toilet) in a comfortable chair

INTERVENTIONS:
Behavioral: Physical activity — Multiple bouts of 3-min brisk walking, every 30 min, for 4 hours.
  Other Names: Walking
  Arms: Walking breaks (WALK)

SUMMARY:
This study will verify the effects of breaking up sitting time with short bouts of light intensity walking on vascular function in women with rheumatoid arthritis.

DETAILED DESCRIPTION:
Women diagnosed with rheumatoid arthritis will participate in this randomized crossover trial. In one of the experimental sessions, the participants will remain 4-h on uninterrupted sitting, and in another day they will perform 3-min light intensity walk every 30 min to break up the sitting position. Vascular function will be assessed before and after each intervention using the following devices/techniques: a) transcranial Doppler ultrasound to assess the middle cerebral artery blood flow velocity at baseline and in response to CO2 breathing (5% CO2 mixture for 3 min), and to repeated sit-to-stand transitions; b) a multi-frequency linear transducer (7-12 MHz) attached to a high-resolution ultrasound machine to assess femoral artery dilation after reactive hyperemia (i.e., flow-mediated dilation); c) a laser Doppler probe attached to the skin surface of the right shin in order to quantify the Laser Doppler flux at baseline and during reactive hyperemia. Additionally, healthy age- and body mass-matched women will be recruited and will only perform the pre-intervention tests.

ELIGIBILITY:
Inclusion Criteria:

* Adult women diagnosed with RA
* From the Rheumatology Clinic at the Liverpool University Hospitals NHS Foundation Trust
* Aged 18-60 yr
* Non-smoker for at least 6months
* Able to provide written informed consent.

Exclusion Criteria:

* Cannot readily read and understand English.
* Currently smoking or within last 6 months.
* Alcohol consumption >14units per week.
* Symptoms of or established cardiovascular disease (except hypertension)
* Previous stroke or myocardial infarction.
* History of diabetes or respiratory disease or chronic kidney disease.
* Musculoskeletal impairment/disability precluding physical activity
* Unstable medication (change in medication within the 3 months)
* Aged <18 or > 60 yr
* Currently pregnant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Middle cerebral artery mean velocity (MCAV) | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  MCAV will be assessed using continuous bilateral transcranial Doppler ultrasound.
Middle cerebral artery mean velocity reactivity to carbon dioxide | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  Participants will breathe a 5% carbon dioxide mixture for 3 min during which time MCAV reactivity to CO2 will be assessed using continuous bilateral transcranial Doppler ultrasound.
Cerebral autoregulation | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  Participants will be asked to complete a series of repeated sit to stand moves (coached by a member of the research team) for a 5-minute period, during which time MCAV will be assessed using continuous bilateral transcranial Doppler ultrasound. Beat by beat blood pressure will also be assessed using finger photoplethysmography.

SECONDARY OUTCOMES:
Brachial artery endothelial function | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  Brachial artery endothelial function will be assessed through flow-mediated dilation using vascular ultrasound.
Finger blood pressure | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  During all procedures, beat by beat finger blood pressure will be measured on the middle finger of the right hand using photoplethysmography.
Superficial femoral artery endothelial function | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  Superficial femoral artery endothelial function will be assessed through flow-mediated dilation using vascular ultrasound.
Skin blood flow response to hyperemia | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  Skin blood flow response to hyperemia will be assessed using a laser doppler probe attached to the shin and forearm.
Stroop color-word test | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  The Stroop color-word test will be implemented to assess attention and inhibitory control.
California Verbal Learning Test-2 | Change from baseline (hour 0) to hour 4 (post-intervention/control)
  Immediate recall of the California Verbal Learning Test-2 will be used to assess verbal learning and memory.
Brachial artery blood flow | Change from baseline to 1-hour/2-hour/3-hour/4-hour
  Vascular ultrasound will be used to assess brachial artery blood flow every hour during the intervention
Femoral artery blood flow | Change from baseline to 1-hour/2-hour/3-hour/4-hour
  Vascular ultrasound will be used to assess femoral artery blood flow every hour during the intervention
Pain intensity | Change from baseline to 1-hour/2-hour/3-hour/4-hour
  Pain intensity will be assessed using a 10cm visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Sport and Exercise Sciences (RISES), Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No